CLINICAL TRIAL: NCT06613867
Title: Wakobo ti Kodro: a Quasi-experimental Study to Improve the Identification and Follow-up of Pregnant Women at Risk of Obstetric Complications in the Community by Traditional Birth Attendants in the Central African Republic
Brief Title: Wakobo-ti-Kodro: Improving Identification of Pregnancy at Risk of Obstetric Complications at Community Level
Status: Completed | Type: Observational
Sponsor: Alliance for International Medical Action (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government); Elrha (Other); PACCI Program (Other)
Responsible Party: Sponsor
Other Study IDs: Wakobo ti Kodro
Record Dates: First submitted 2024-09-19; First posted 2024-09-26 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Maternal Health; Pregnancy Complications
Keywords: Traditional birth attendant; Digital health; Pregnancy at risk of complications identification; Collaboration with traditional birth attendant; Africa; Central African Republic
MeSH Terms: conditions — Pregnancy Complications

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Wakobotikodro — Wakobotikodro : an intervention combining (i) training matrons to identify and monitor high-risk pregnancies, (ii) integrating them into the healthcare system and (iii) using a digital decision-support application installed on a smartphone and adapted to their profile, could improve the identification and monitoring of high-risk pregnancies.

SUMMARY:
This project aims to improve maternal health indicators in a national context where the maternal mortality rate is one of the highest in the world. Our hypothesis is that an intervention combining (i) the training of traditional birth attendant in the identification and monitoring of high-risk pregnancies, (ii) their integration into the health system and (iii) the use of a digital decision-support application installed on a smartphone and adapted to their profile, could strengthen the identification and monitoring of high-risk pregnancies, increase attendance at facilities and thus the rate of assisted deliveries in health facilities, in Bimbo district around the capital Bangui in the Central African republic.

DETAILED DESCRIPTION:
This is a quasi-experimental study with a before (baseline measurement) and after (final measurement) approach combined with 2) an exploratory prospective observational cohort study and 3) a sub-study using a mixed methodology.

The main objective is to assess a composite intervention implementation combining the integration of Traditional Birth Attendants (TBAs) into the health system through a strengthened collaboration with health facilities with the support of a numeric application aiming at registering pregnant women & identifying those at high risk of obstetric complications.

The secondary objectives are to:

1. Describe the characteristics of antenatal care, pregnancy outcomes, postnatal care, maternal and neonatal mortality, and changes in the use of health facilities by pregnant women.
2. To assess the acceptability and feasibility of this intervention with matrons, community health workers, community representatives, women who have already given birth in the study area and health staff involved in the study, in order to understand the potential levers and barriers to the implementation of the intervention.

ELIGIBILITY:
Inclusion Criteria for the main study (quasi-experimental study with a before-after approach)

* Aggregated data of pregnant women, regardless of the age of their pregnancy, and
* attending the health facilities included in the study

Inclusion Criteria for participating in the observational cohort:

* Being a pregnant woman residing in the study area and
* attending the health facilities included in the study and
* with a given individual consent.

Inclusion Criteria for participating in the sub-study on intervention's acceptability and feasibility:

* traditional birth attendants (TBAs) or
* health workers working in health facilities or
* community health workers or
* community representatives or
* women who have already given birth or pregnant women or their husbands AND
* All with a given individual consent AND
* All being part of the study area.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The main study population is pregnant women attending the health facilities included in the study.
  Secondary population are beneficiaries of the intervention tested: traditional birth attendants, health workers, community health workers, community representatives, women who have already given birth or pregnant women or their husbands living in the study area.
Sampling Method: Non-Probability Sample
Enrollment: 1857 (Actual)
Dates: Start 2023-07-17 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Deliveries in health facilities of women with complicated pregnancies | Comparison between baseline and endline data after 10 months of intervention
  Proportion of deliveries by pregnant women at risk of obstetric complications among all women who give birth in the health facilities included in the study, after 10 months of intervention

SECONDARY OUTCOMES:
Antenatal consultancies (ANCs) | after 10 months of intervention
  Evolution of monthly number of ANCs at health facilities
Delivery | after 10 months of intervention
  Evolution of monthly number of delivery at health facilities
Post-partum consultancies | after 10 months of intervention
  Evolution of monthly number of Post-partum consultancies at health facilities
Pregnant women at risk of obstetrical complication, screened by traditional birth attendants in the community | after 10 months of intervention
  Evolution of monthly number of Pregnant women at risk, screened by traditional birth attendants in the community
Pregnant women at risk of obstetrical complication, monitored at health facilities | after 10 months of intervention
  Evolution of monthly number of Pregnant women at risk of obstetrical complication, monitored at health facilities
Maternal mortality rate | after 10 months of intervention
  Number of death of women while pregnant or within 42 days of termination of pregnancy
Neonatal mortality rate | after 10 months of intervention
  Death of a live born infant, regardless of gestational age at birth, within the first 28 completed days of life

CONTACTS AND LOCATIONS:
Overall Officials: Richard Ngbale, Pr, Principal Investigator — Faculté des sciences de la santé, Bangui; Renaud Becquet, Principal Investigator — Institut National de la Santé Et de la Recherche Médicale, France
Locations (1):
- Bimbo health center,, Bimbo, Bangui Prefecture, Central African Republic

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: web page of Inserm website — https://www.bordeaux-population-health.center/fr/video-wakobo-ti-kodro-ameliorer-grossesses-risque-republique-centrafricaine/
- See also: page web of ELRHA website — https://www.elrha.org/project/nassamba/